CLINICAL TRIAL: NCT03183297
Title: A Double-Blind, Placebo-Controlled, 4-Way Crossover Study to Evaluate the Pharmacokinetics and Pharmacodynamics at Two Dose Levels of JMI-001 in Comparison With Fexofenadine and Naproxen Administered in Conjunction With Alcohol.
Brief Title: Study to Evaluate the Pharmacokinetics and Pharmacodynamics of JMI-001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sen-Jam Pharmaceutical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SJP-1-01
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Veisalgia
MeSH Terms: interventions — Naproxen; fexofenadine

STUDY DESIGN:
Intervention Model Description: A Double-Blind, Placebo-Controlled, 4-Way Crossover Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JMI-001 (Experimental): JMI-001 is a combination product of naproxen 220mg and fexofenadine 60mg (Dose Level one) then a combination product of naproxen 440mg and fexofenadine 120mg (Dose Level Two).
  Interventions: Drug: JMI-001
- Naproxen (Active Comparator): Naproxen 220mg or 440mg
  Interventions: Drug: Naproxen; Drug: placebo
- Fexofenadine (Active Comparator): fexofenadine 60mg or 120mg
  Interventions: Drug: Fexofenadine; Drug: placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: JMI-001 — JMI-001, a combination product of naproxen and fexofenadine
  Arms: JMI-001
Drug: Naproxen — Naproxen sodium 220mg
  Arms: Naproxen
Drug: Fexofenadine — Fexofenadine 60mg
  Arms: Fexofenadine
Drug: placebo — placebo comparator
  Arms: Fexofenadine; Naproxen; Placebo

SUMMARY:
This will be a double-blind, placebo-controlled study with a 4-way crossover design with subjects administered study drug (JMI-001), placebo, fexofenadine alone and naproxen alone on different study days, in conjunction with a quantity of alcohol estimated to be sufficient to produce a hangover the next day. The primary objective of the study is the evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of two different doses of JMI-001 administered in conjunction with alcohol to healthy adult subjects.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled study with a 4-way crossover design with subjects administered study drug (JMI-001), placebo, fexofenadine alone and naproxen alone on different study days, in conjunction with a quantity of alcohol estimated to be sufficient to produce a hangover the next day. The primary objective of the study is the evaluate the pharmacokinetics and pharmacodynamics of two different doses of JMI-001 administered in conjunction with alcohol to healthy adult subjects. The secondary objective of this study is to compare the PK characteristics of fexofenadine administered as JMI-001 with administration of fexofenadine alone, and the PK characteristics of naproxen administered as JMI-001 with administration of naproxen alone. To compare overall hangover severity after administering JMI-001 with overall hangover severity after administration of fexofenadine alone or naproxen alone. To analyze possible quantitative differences in symptom profiles by treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking men or women between 21 and 65 years inclusive; 2. Good general health as determined by a thorough medical history and physical examination including vital signs; 3. Subject is a self-reported moderate drinker of alcohol, typically consuming 2 to 7 units of alcohol. Moderate drinking can be approximated with a BAC of 0.04 - 0.11%. The 0.04% - 0.11% BAC correlates approximately with a 120-160 pound female drinking 2 to 5 drinks in 2 to 3 hours, respectively, and a 160-200 pound male drinking 3 to 7 drinks in 2 to 3 hours, respectively; 4. Subject has prequalified as likely hangover-sensitive based on pre-study questionnaire; 5. Body mass index between 19 and 32 kg/m2, inclusive ; 6. Report a regular, habitual bedtime between 21:30 and 24:00; 7. Females of childbearing potential must have a negative urine pregnancy test at screening and upon admission for each treatment visit and be using an acceptable method of contraception (see Section 8.5); 8. Subject is capable of understanding the requirements of the study and to give written informed consent; 9. Subject is able to follow study instructions and is willing to complete all study visits and procedures.

-

Exclusion Criteria:

1. Acute illness within 14 days prior to screening visit; 2. Allergic reaction or upper respiratory tract infection within 7 days of screening visit; 3. Vaccination administration within 7 days of screening visit; 4. Clinically significant, unstable medical illness; 5. Evidence or history of clinically significant autoimmune, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic or neurological disease; 6. History of cancer or diabetes; 7. Subject has a previous or current Substance-Related Disorder as defined by DSM 5; 8. A score of 8 or greater on the AUDIT scale; 9. Self-report of recent (within one month) or current use of smoked or chewed tobacco products, or use of nicotine (e.g., nicotine gum or patch); 10. Positive alcohol Breathalyzer test at check-in for any treatment visit; 11. Positive urine drug screen at screening or at check-in for any treatment visit; 12. A seated blood pressure > 140/90 mm/Hg at screening; 13. Heart rate > 100 beats per minute at screening; 14. Subjects who are unwilling to forgo caffeine consumption with or following dinner on each treatment night or who are unwilling to comply with study restrictions for prohibited medications/ foods throughout study participation; 15. Clinically significant psychiatric illness, including chronic psychiatric illness or the history or presence of any Axis I condition; 16. Any clinically significant abnormal finding on physical examination or vital signs; 17. Subject has previously experienced an allergic reaction or adverse event associated with aspirin, NSAIDs, or antihistamine usage; 18. Subject requires the use of any prescription or over-the-counter (OTC) oral pain medication(s) on study treatment days; 19. Women who are breastfeeding; 20. Any medical condition or any condition or situation that in the investigator's opinion may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study; 21. Concurrent participation in an investigational drug or device study, or use of any investigational drug within 30 days prior to screening.

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 24 hours
  Maximum Plasma Concentration of each drug measured in ng/mL
Time to Maximum Plasma Concentration (Tmax) | 24 hours
  Time to achieve the (Cmax) for each drug measured in hours
Area Under the Curve (AUC) | 24 hours
  Area Under the Curve for each drug measured in h*ng/mL
Elimination half-life | 24 hours
  Elimination half-life measured in hours

SECONDARY OUTCOMES:
Hangover Severity Score | 24 hours
  Single item Hangover Score subjectively measured by the subject from 0=no symptoms to 10=worst symptoms
Multiple Symptom Hangover Severity Score | 24 hours
  A composite score derived from a spectrum of hangover symptoms (23-items) with each symptom subjectively measured by the subject from 0=no symptom to 10=worst symptom

CONTACTS AND LOCATIONS:
Overall Officials: Magdy L Shenouda, MD, Principal Investigator — Clinilabs, Inc.

IPD SHARING:
Plan to Share IPD: No